CLINICAL TRIAL: NCT06967532
Title: Efficacy of Torque Teno Virus as a Biomarker for Predicting Treatment Response of Immune Checkpoint Inhibitor Therapy and Postoperative Outcome in NSCLC Patients - A Prospective Non-interventional Single-arm Study
Brief Title: Efficacy of Torque Teno Virus as a Biomarker for Predicting Treatment Response of Immune Checkpoint Inhibitor Therapy and Postoperative Outcome in NSCLC Patients
Acronym: TTV in NSCLC
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Aigner, Professor of Thoracic Surgery, Medical University of Vienna
Other Study IDs: 1619/2024
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — Blood sampling

SUMMARY:
First discovered in 1997 the torque teno virus (TTV) can be found in the vast majority of the human population throughout their lifetime. The TTV levels correlate with infectious diseases and organ rejection and are therefore currently being investigated as a tool to optimize the management of patients after solid organ transplantation (SOT). While TTV levels are already tested to guide immunosuppressive therapy its significance for oncologic patients is unclear. In recent years immune checkpoint inhibitors (ICIs) are increasingly implemented in multimodal therapy approaches for patients with non-small-cell lung cancer (NSCLC). Since ICI and TTV levels depend on T-cell function, the TTV load may be a relevant biomarker for the treatment response as well as complication risk after ICI therapy. Current standard imaging using PERCIST and RECIST criteria is prone to misinterpretation of treatment response of ICI therapy due to pseudoprogression and nodal immune flaring. This study aims to prospectively analyze TTV levels in NSCLC patients before, during and after neoadjuvant chemo-immunotherapy and correlate inter- and intraindividual changes in TTV levels with response rates observed on PET/CT restaging and histopathological response rates as well as postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

- Histologically or cytologically verified NSCLC stage II-IV (OMD) according to UICC TNM8 edition considered operable in curative intent after neoadjuvant systemic therapy containing immune checkpoint inhibition by local multidisciplinary tumor board (MDT) decision.

ECOG < or = 1 Staging with PET/CT and cMRI/CCT Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged > 18 years. Women of childbearing potential are eligible and must provide a negative serum or urine pregnancy test and follow instructions for contraception.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Histopathological response to neoadjuvant chemo-immunotherapy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with scientific institutions upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF